CLINICAL TRIAL: NCT00560287
Title: Role of Non-invasive Ventilation in Amyotrophic Lateral Sclerosis: Volume Versus Pressure Mode
Brief Title: Non-Invasive Ventilation in Amyotrophic Lateral Sclerosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Salvatore Maugeri (Other)
Responsible Party: Stefano Nava, Fondazione S.Maugerii
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 190H09; 190H09
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Last update posted 2010-03-29 (Estimated); Status verified 2010-03

CONDITIONS: Amyotrophic Lateral Sclerosis; Chronic Respiratory Failure
Keywords: Amyotrophic Lateral Sclerosis; Non-invasive ventilation; Chronic Respiratory Failure
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Volume assist non-invasive ventilation
  Interventions: Device: Non invasive ventilation delivered with one of the ventilator specifically designed for NIV and given to the patient by the home care providers; Device: Non invasive ventilation
- 2 (Active Comparator): Pressure Assist mode
  Interventions: Device: Non invasive ventilation delivered with one of the ventilator specifically designed for NIV and given to the patient by the home care providers; Device: Non invasive ventilation

INTERVENTIONS:
Device: Non invasive ventilation delivered with one of the ventilator specifically designed for NIV and given to the patient by the home care providers — A very recent randomized controlled trial show that in ALS without severe bulbar dysfunction, NIV improves survival with maintenance of, and improvement in, quality of life, including sleep quality. The survival benefit from NIV in this group is much greater than that from currently available neuroprotective therapy, like riluzole.
  Other Names: Legendaire (Airox); Vivo (Breas); Elisee (Saime); Synchrony (Respironics)
Device: Non invasive ventilation — A very recent randomized controlled trial show that in ALS without severe bulbar dysfunction, NIV improves survival with maintenance of, and improvement in, quality of life, including sleep quality. The survival benefit from NIV in this group is much greater than that from currently available neuroprotective therapy, like riluzole.
  Other Names: Legendaire (Airox); Vivo (Breas); Elisee (Saime); Synchrony (Respironics)

SUMMARY:
Non-invasive mechanical ventilation (NIV) has been increasingly used as a treatment of chronic hypercapnic respiratory failure. Its use in patients affected by chronic obstructive pulmonary disorders is still controversial, while most of the studies performed in restrictive thoracic disorders (RTD), and in particular in neuromuscular patients, suggested alleviation of the symptoms of chronic hypoventilation in the short term, and in two small studies survival was prolonged.

In the terminal phase of the disease, when the respiratory muscles became weaker it is very likely that the operators need to frequently adjust the level of inspiratory pressure in an attempt to guarantee an adequate tidal volume, so that alveolar hypoventilation may be avoided.

Theoretically the use of a volume assisted ventilation may overpass this problem of frequent variations of the settings, since the provision of a fixed tidal volume may always guarantee and adequate alveolar ventilation.

The primary aims of this multicenter randomized study are to evaluate the clinical efficacy, the patients' tolerance and quality of life and the frequency of changing settings in a group of patients with SLS and initial chronic respiratory failure undergoing long-term NIV with Pressure Support Ventilation or Volume Assisted Ventilation.

DETAILED DESCRIPTION:
Background

Non-invasive mechanical ventilation (NIV) has been increasingly used as a treatment of chronic hypercapnic respiratory failure. Its use in patients affected by chronic obstructive pulmonary disorders is still controversial, while most of the studies performed in restrictive thoracic disorders (RTD), and in particular in neuromuscular patients, suggested alleviation of the symptoms of chronic hypoventilation in the short term, and in two small studies survival was prolonged. As a matter of fact a recent Cochrane review stated that "long-term mechanical ventilation should be offered as a therapeutic option to patients with chronic respiratory failure due to neuromuscular diseases". Recurrent episodes of nocturnal desaturation especially during REM sleep may deeply influence the prognosis of patients affect by these disorders (i.e. ALS), and they are often associated with hypercapnia, so that the correction of nocturnal hypoventilation seems to be the major goal to achieve with the ventilatory treatment.

A very recent randomized controlled trial show that in ALS without severe bulbar dysfunction, NIV improves survival with maintenance of, and improvement in, quality of life, including sleep quality. The survival benefit from NIV in this group is much greater than that from currently available neuroprotective therapy, like riluzole.

Most of the studies performed in RTD disorders were performed using a pressure assisted mode (i.e Pressure Support Ventilation), because of the supposed better tolerance of the patients and easy of settings for the operators, even though this has never been scientifically proven.

In the terminal phase of the disease, when the respiratory muscles became weaker it is very likely that the operators need to frequently adjust the level of inspiratory pressure in an attempt to guarantee an adequate tidal volume, so that alveolar hypoventilation may be avoided.

Theoretically the use of a volume assisted ventilation may overpass this problem of frequent variations of the settings, since the provision of a fixed tidal volume may always guarantee and adequate alveolar ventilation.

The primary aims of this multicenter randomized study are to evaluate the clinical efficacy, the patients' tolerance and quality of life and the frequency of changing settings in a group of patients with SLS and initial chronic respiratory failure undergoing long-term NIV with Pressure Support Ventilation or Volume Assisted Ventilation.

Aim of the Project

The primary aims of the project are to evaluate the clinical efficacy, the patients' tolerance and quality of life and the frequency of changing settings in a group of patients with SLS and initial chronic respiratory failure undergoing long-term NIV with Pressure Support Ventilation or Volume Assisted Ventilation.

• Enrollment criteria: Patients with the diagnosis of ALS and one of the following signs: 1) Vital Capacity < 50% predicted 2) a Maximal Inspiratory Pressure (MIP) < 60% predicted 3) polygraphic signs of nocturnal hypoventilation with daytime symptoms.

- The patients will be randomized to receive NIV with one of the following modes: 1) Pressure Support Ventilation with the inspiratory pressure set according to the patient's tolerance in order to achieve an expired tidal volume > 6 ml/Kg and <8ml/Kg. The back-up rate will be set at 10 breaths/min. 2) Volume assist ventilation with a back-up rate of 10 breaths/min and a tidal volume set to achieve an expired tidal volume > 6 ml/Kg and <8ml/Kg

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of ALS and one of the following signs:

  * Vital Capacity < 50% predicted
  * A Maximal Inspiratory Pressure (MIP) < 60% predicted
  * Polygraphic signs of nocturnal hypoventilation with daytime symptoms.

Exclusion Criteria:

* Life expectancy>12 months
* Any comorbidity
* Acute Respiratory Failure

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-08 (Actual); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
quality of life | 1 year
tolerance to NIV | 1 year
number of hours of NIV per day | 1 year
frequency of hospital admission | 1 year
frequency of changing the ventilator settings by the operator. | 1 year

SECONDARY OUTCOMES:
survival | 1 year
diurnal and nocturnal gas exchange | 1 year
Pulmonary Function Tests (PFTs). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Nava, Principal Investigator — Fondazione Salvatore Maugeri; Stefano Nava, MD, Principal Investigator — Fondazione S.maugeri
Locations (2):
- Italy (2):
  - Fondazione S.Maugeri, Pavia
  - Respiratory Unit FSM, Pavia